CLINICAL TRIAL: NCT03923270
Title: Sequential Maintenance With Thoracic Radiotherapy and Durvalumab (MEDI4736) Monotherapy or Durvalumab (MEDI 4736) Combinations (Tremelimumab or Olaparib) in Patients With Extensive Stage-Small Cell Lung Cancer After First Line Platinum Based Chemotherapy
Brief Title: Radiotherapy and Durvalumab/Durvalumab Combo (Tremelimumab/Olaparid) for Small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-19942
Record Dates: First submitted 2019-03-11; First posted 2019-04-22 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Small Cell Lung Cancer Extensive Stage; Small-cell Lung Cancer
Keywords: lung cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma; Lung Neoplasms | interventions — durvalumab; tremelimumab; olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Thoracic Radiotherapy plus Durvalumab (No Intervention): This Arm is a standard of care Arm. Patients will receive thoracic radiotherapy (30 Gray units total, 3 Gray units X 10 fractions), then in 2-3 weeks begin 1500 mg intravenously of Durvalumab every 4 weeks for up to 13 doses
- Thoracic Radiotherapy plus Durvalumab and 75mg Tremelimumab (Experimental): Patients will receive thoracic radiotherapy (30 Gray units total, 3 Gray units X 10 fractions), then in 2-3 weeks begin 1500 mg intravenously of Durvalumab every 4 weeks for up to 4 doses and 75mg intravenously of Tremelimumab every 4 weeks for up to 4 doses
  Interventions: Drug: Durvalumab; Drug: Tremelimumab; Radiation: Thoracic Radiotherapy
- Thoracic Radiotherapy plus Durvalumab and Olaparib (Experimental): Patients will receive thoracic radiotherapy (30 Gray units total, 3 Gray units X 10 fractions), then in 2-3 weeks begin 1500 mg intravenously of Durvalumab every 4 weeks and 300 mg orally of Olaparib twice a day
  Interventions: Drug: Durvalumab; Drug: Olaparib Pill; Radiation: Thoracic Radiotherapy
- Thoracic Radiotherapy plus Durvalumab and 300mg Tremelimumab (Experimental): Patients will receive thoracic radiotherapy (30 Gray units total, 3 Gray units X 10 fractions), then in 2-3 weeks begin 1500 mg intravenously of Durvalumab every 4 weeks and 300 mg Tremelimumab IV x 1 (single dose)
  Interventions: Drug: Durvalumab; Radiation: Thoracic Radiotherapy; Drug: Tremelimumab

INTERVENTIONS:
Drug: Durvalumab — Participants in all arms will be administered 1500 mg of Durvalumab intravenously every 4 weeks.
  Other Names: Imfinzi; MEDI4736
  Arms: Thoracic Radiotherapy plus Durvalumab and 300mg Tremelimumab; Thoracic Radiotherapy plus Durvalumab and 75mg Tremelimumab; Thoracic Radiotherapy plus Durvalumab and Olaparib
Drug: Tremelimumab — Participants in arm B will be administered 75 mg of Tremelimumab intravenously every 4 weeks for up to 4 doses.
  Arms: Thoracic Radiotherapy plus Durvalumab and 75mg Tremelimumab
Drug: Olaparib Pill — Participants in arm C will be self-administer 300 mg of Olaparib orally.
  Other Names: Lynparza; MK-7339
  Arms: Thoracic Radiotherapy plus Durvalumab and Olaparib
Radiation: Thoracic Radiotherapy — Thoracic Radiotherapy will be administered at 3 Gray units X 10 fractions
  Arms: Thoracic Radiotherapy plus Durvalumab and 300mg Tremelimumab; Thoracic Radiotherapy plus Durvalumab and 75mg Tremelimumab; Thoracic Radiotherapy plus Durvalumab and Olaparib
Drug: Tremelimumab — Participants in arm D will be administered 300 mg of Tremelimumab intravenously in 1 single dose
  Arms: Thoracic Radiotherapy plus Durvalumab and 300mg Tremelimumab

SUMMARY:
This is a randomized multi-arm trial evaluating the safety and efficacy of thoracic radiation therapy followed by either durvalumab as monotherapy or in combination with tremelimumab or olaparib in participants with Extensive-Stage Disease Small Cell Lung Cancer (ES-SCLC) who have completed a first-line platinum-based chemotherapy regimen and achieved ongoing complete response (CR), partial response (PR) or stable disease (SD).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Body weight greater than 30 kg
* Participants must be willing and able to comply with scheduled visits, treatment schedule, laboratory tests and other requirements of the study.
* Participants must have small cell lung cancer, documented by histology or cytology from brushing, washing, fine needle aspiration or core biopsy from a defined lesion, but not from sputum cytology alone. No mixed histologies allowed.
* Participants must be presented at initial diagnosis with extensive-stage disease (ES-SCLC).
* Eastern Cooperative Oncology Group (ECOG) Performance status 0 or 1.
* Participants must have received 4-6 cycles of platinum-based first-line chemotherapy and must have an ongoing complete response (CR), partial response (PR), or stable disease (SD) after completion. Acceptable combinations (NCCN guidelines), include cisplatin or carboplatin with etoposide or irinotecan. As an exception to the above criterion, participants receiving only 3 cycles of chemotherapy due to toxicity are eligible, if they have an ongoing PR or CR after the 3rd cycle. Participants who have received > 6 cycles of platinum-based first-line chemotherapy are not eligible. Participants receiving checkpoint inhibitor (CPI) monotherapy (anti-PD-1, anti-PD-L1, others) as part of their first line chemotherapy treatment will be eligible as long as they discontinue the CPI prior to the start of thoracic radiotherapy.
* Participants must initiate study treatment with thoracic XRT ≤ 60 days from the last dose of platinum- based first line chemotherapy;
* Whenever possible, a formalin-fixed, paraffin-embedded (FFPE) tumor tissue block or 5-10 unstained slides of tumor sample (archival) should be made available (less material is acceptable);
* Participants must have a life expectancy of 16 weeks or more.
* Active infection including: tuberculosis, hepatitis B (known positive hepatitis B surface antigen (HBsAg) result) and/or, hepatitis C. Patients with a past or resolved hepatitis B infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA (indicating no current infection).
* Known positive test for human immunodeficiency virus (positive HIV 1/2 antibodies) or known medical history of acquired immunodeficiency syndrome (AIDS)
* Adequate bone marrow function measured within 28 days prior to administration of study as defined per protocol.
* Adequate rental function as defined per protocol.
* Adequate hepatic function as defined per protocol
* Women of childbearing potential (WOCBP) patients or male patients who are sexually active with WOCBP and female partners of male participants must agree to follow instructions of "highly effective methods of contraception) per protocol for duration of treatment with study drug(s) plus the specified washout period.
* Male participants must be willing to refrain from sperm donation during the study and for at least 180 days after the last dose of durvalumab combination therapy, 90 days after the last dose of durvalumab or olaparib monotherapy.

Exclusion Criteria:

* Participants with previous brain metastases are eligible provided that they are treated, are asymptomatic, and have stable disease at the screening tumor assessment. A ≥ 2 week disease stable interval as confirmed by MRI or CT brain w/ contrast (Table 7.4-2) is required after treatment of brain metastases before initiation of thoracic XRT. In addition, subjects must have been either off corticosteroids, or on a stable or decreasing dose of ≤10 mg daily prednisone (or equivalent).
* Participants who have received prior thoracic XRT are excluded.
* Participants with Carcinomatous meningitis
* Pregnant or breastfeeding women
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease, systemic lupus erythematosus, rheumatoid arthritis, Wegener syndrome and hypophysitis or uveitis. Patients with an autoimmune paraneoplastic syndrome requiring concurrent immunosuppressive treatment are excluded. Patients with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll
* Participants with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of study treatment (excluding thoracic radiotherapy). Some exceptions apply.
* Prior CPI therapy with anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody (including any other antibody or drug specifically targeting T cell co-stimulation or checkpoint pathways). Exception: CPI use with first line chemotherapy that is stopped prior to trial enrollment.
* Participants who have received any previous treatment with a Poly ADP Ribose Polymerase (PARP) inhibitor, including olaparib
* Interstitial lung disease (ILD): Any evidence of current ILD or pneumonitis or a prior history of ILD or pneumonitis requiring oral or IV glucocorticoids.
* Previous malignancies unless a complete control (no evidence of disease) was achieved ≥ 2 years prior to study entry AND no additional therapy is required during the study period (EXCEPT: adequately treated non-melanoma skin cancer, curatively treated in situ cancer and stage 1, grade 1 endometrial cancer).
* Participants with a known medical condition that, in the investigator's opinion, would increase the risk associated with study participation or study drug(s) administration or interfere with the interpretation of safety results.
* Major surgery or significant traumatic injury that is not recovered at least 14 days before the initiation of thoracic radiation therapy
* All toxicities attributed to prior anti-cancer therapy must have been resolved to Grade 1 (NCI CTCAE Version 5.0) or baseline before administration of study drug(s). Some exceptions apply.
* Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
* Patients with known contraindications to radiotherapy, including inherited syndromes associated with hypersensitivity to ionizing radiation (e.g., Ataxia-Telangiectasia, Nijmegen Breakage Syndrome).
* History of allergy or hypersensitivity to any of the study drugs or study drug components

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-06-06 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Unacceptable Serious Adverse Events (SAEs) | 13 weeks
  Unacceptable toxicity status at the end of 13-week safety observation period with unacceptable toxicity defined as:
  * Any grade 4 immune related adverse event (irAE),
  * Any ≥ grade 3 noninfectious pneumonitis,
  * Any ≥ grade 3 colitis,
  * Any grade 3 irAE, excluding colitis or pneumonitis, that does not downgrade to grade 2 within 7 days after onset of the event despite optimal medical management including systemic corticosteroids or does not downgrade to ≤ grade 1 or baseline within 14 days,
  * Liver transaminase elevation > 8 × Upper Limit of Normal (ULN) or total bilirubin > 5 × ULN
  * Any ≥ grade 3 non-irAE with exceptions per protocol
Phase IB: Progression Free Survival | 6 months
  Progression Free Survival (PFS) defined as the duration from date of registration to date of first documentation of progression assessed by local investigator or symptomatic deterioration or death due to any cause. Patients last known to be alive are censored at date of last contact.

SECONDARY OUTCOMES:
Median Progression Free Survival | Up to 12 months
  Progression Free Survival (PFS) is defined as the duration from date of registration to date of first documentation of progression assessed by local investigator or symptomatic deterioration (as defined above) or death due to any cause. Patients last known to be alive are censored at date of last contact.
Overall Survival | Up to 12 months
  Overall Survival (OS) will is defined as the duration from date of registration to date of death due to any cause. Patients last known to be alive are censored at date of last contact.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto A Chiappori, MD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No